CLINICAL TRIAL: NCT04631926
Title: The Impact of Hip Exercises on Pelvic Floor Muscle Strength and Function as a Potential Non-surgical Management for Urinary Incontinence in Older Women
Brief Title: The Impact of Hip Exercises on Pelvic Floor Muscle Strength and Function in Older Women With Urinary Incontinence
Acronym: WIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Isuzu Meyer, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Women & Urinary INcontinence
Record Dates: First submitted 2020-11-06; First posted 2020-11-17 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Urinary Incontinence; Geriatric Syndrome
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hip Muscle Exercises (Other): Hip Muscle Exercises
  Interventions: Behavioral: Hip Muscle Exercise

INTERVENTIONS:
Behavioral: Hip Muscle Exercise — Standardized 12-week hip muscle exercises focusing on the external hip rotators with progressive resistance

SUMMARY:
This is a prospective cohort study of 30 older women ages 65 and older with urinary incontinence (UI) who will under go a standardized 12-week hip muscle exercises (isometric strengthening of hip external rotators with progressive resistance training).

DETAILED DESCRIPTION:
This is a prospective cohort study of 30 older women ages 65 and older with urinary incontinence (UI) who will under go a standardized 12-week hip muscle exercises (isometric strengthening of hip external rotators with progressive resistance training). Participants will take part in a 12-week hip muscle exercise program (weekly supervised hip exercises with resistance progression) plus a home program with the same exercises 3 days per week. the exercise program will be administered by the licensed physical therapist with special focus in hip strength. The change in pelvic floor muscle strength (peak pelvic floor muscle squeeze pressures) pre- to post hip muscle exercises. Changes in UI symptom severity, and impact of UI symptoms on quality of life will be assessed. Objective measurement of pelvic floor muscle strength will be obtained using a perineometer. UI symptom severity and quality of life will be measured using validated questionnaires (PFDI and PFIQ, respectively).

ELIGIBILITY:
Inclusion Criteria:

* Women ages ≥65
* UI for at least the last 3 months UI will be defined using the following (a widely-accepted definition in epidemiologic studies) Scores 3 - 12 on the validated 2-item Incontinence Severity Index (ISI)

Exclusion Criteria:

* Women unable to follow-up, not willing to, or unable to participate in the exercise intervention program
* Prior or current treatment for UI including previous FDA approved medications for UI, prior surgery for UI within the past 12 months
* Pelvic organ prolapse beyond the hymen
* Potential causes or conditions associated with neurogenic bladder (multiple sclerosis, Parkinson's disease, stroke, spinal cord injury)
* Urinary retention, incomplete bladder emptying (via bladder scan, >150mL post-void residual)
* Conditions (neurological or musculoskeletal) that compromise mobility, requiring assisted device for ambulation or wheel chair
* Diagnosis of dementia or cognitive impairment (Montreal Cognitive Assessment [MoCA] <25, mild cognitive impairment)

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — 65 and older
Enrollment: 32 (Actual)
Dates: Start 2022-02-21 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Pelvic floor muscle strength | Baseline
  pelvic floor muscle strength (peak pelvic floor muscle squeeze pressures) pre hip muscle exercises
Pelvic floor muscle strength | 12 weeks
  pelvic floor muscle strength (peak pelvic floor muscle squeeze pressures) post hip muscle exercises

SECONDARY OUTCOMES:
Urinary incontinence symptom severity | Baseline
  urinary incontinence specific symptom severity - Validated questionnaire score Pelvic Floor Disability Index (PFDI), pre hip muscle exercises. PFDI Questionnaire is for certain bowel, bladder, or pelvic symptoms and, see, how much they bother. The PFDI-20 has 20 items and 3 scales of your symptoms. All items use the following format with a response scale from 0 not present to 4 worst. Symptom scale: 0 = not present 1= not at all 2 = somewhat 3 = moderately 4 = quite a bit
Urinary incontinence symptom severity | 12 weeks
  urinary incontinence specific symptom severity - Pelvic Floor Disability Index (PFDI), post hip muscle exercises. PFDI Questionnaire is for certain bowel, bladder, or pelvic symptoms and, see, how much they bother. The PFDI-20 has 20 items and 3 scales of your symptoms. All items use the following format with a response scale from 0 not present to 4 worst. Symptom scale: 0 = not present 1= not at all 2 = somewhat 3 = moderately 4 = quite a bit
Impact of urinary incontinence symptoms on quality of life | Baseline
  impact of urinary incontinence symptoms on quality of life - validated questionnaire score Pelvic Floor Impact Questionnaire (PFIQ), pre muscle exercises. It is a health-related quality of life questionnaire for women with pelvic floor conditions. PFIQ has 7 questions and each question has 3 separate responses (one for each of 3 scales). All of the items use the following response scale: 0 = Not at all; 1 = Somewhat; 2 = Moderately; 3 = Quite a bit Scales:
Impact of urinary incontinence symptoms on quality of life | 12 weeks
  impact of urinary incontinence symptoms on quality of life - validated questionnaire score (PFIQ), post muscle exercises. It is a health-related quality of life questionnaire for women with pelvic floor conditions. PFIQ has 7 questions and each question has 3 separate responses (one for each of 3 scales). All of the items use the following response scale: 0 = Not at all; 1 = Somewhat; 2 = Moderately; 3 = Quite a bit Scales:

CONTACTS AND LOCATIONS:
Overall Officials: Isuzu Meyer, MD. MSPH, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Kirklin Clinic of Uab Hospital, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No